CLINICAL TRIAL: NCT04235504
Title: ADvanced Hybrid Closed Loop Study in Adult Population With Type 1 Diabetes
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP327
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Type 1 Diabetes
Keywords: Advanced Hybrid Closed Loop; Multiple Daily Injections; Flash Glucose Monitoring; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: There will be 2 Cohort for this study:
  1. Cohort A: Subjects on MDI + FGM will be randomized into: Treatment Arm (AHCL) and Control Arm (MDI+ FGM)
  2. Cohort B: Subjects on MDI + Real-Time CGM will be randomized into: Treatment Arm (AHCL) and Control Arm (MDI+ CGM) (exploratory analysis)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Control Arm (Active Comparator): The Control Arm will use individual subject's current diabetes therapy (MDI+FGM or MDI+CGM) for 6 months during the Study Phase. During the Continuation Phase of 6 months Control Arm will start using the Advance Hybrid Close Loop (AHCL) MiniMed™ 670G system version 4.0
  Interventions: Other: MDI; Device: AHCL
- Treatment Arm (Experimental): The Treatment Arm will use the Advance Hybrid Close Loop (AHCL) MiniMed™ 670G system version 4.0 for 6 months during the Study Phase and other 6 months during the Continuation Phase.
  Interventions: Device: AHCL

INTERVENTIONS:
Other: MDI — Subject continues their standard Multiple Daily Injections therapy with FGM or RT-CGM
  Arms: Control Arm
Device: AHCL — Subject starts using the Advance Hybrid Close Loop (AHCL) MiniMed™ 670G system version 4.0.
  Starting time depends on which Arm the subject is assigned to: if the subject is assigned to the Treatment Arm, then the intervention starts after the RUN-IN period. If the subject is assigned to the Control Arm the intervention will start after 6 months from the date of the enrollment.

SUMMARY:
The purpose of this study evaluate the safety and efficacy of the Advanced Hybrid Closed Loop (AHCL) system in sub-optimally controlled patients with T1D, in comparison with Multiple Daily Injection (MDI) therapy with Flash Glucose Monitoring (FGM) or Continuous Glucose Monitoring (CGM). Patient with a diagnosis of Type 1 diabetes currently under MDI+ FGM or MDI+ CGM therapy will be enrolled.

DETAILED DESCRIPTION:
This study is a pre-market, multi-center, prospective, open label, adaptative, randomized controlled trial in insulin-requiring adult subjects with type 1 diabetes on MDI therapy. The study will have three period:

1. Run-in Phase: The Run-in period is of 4 weeks (and can be extended for 2 additional ones) during which time a blinded CGM sensor will be worn for two weeks.
2. Study Phase: There will be a 6 months randomized study period with two arms: Treatment Arm (AHCL) and the Control Arm.
3. Continuation Phase: There will be a 6 months continuation phase during which time all the subjects will use the AHCL system.

Approximately 124 subjects will be enrolled in the study up to 20 investigational centers in EMEA.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is age ≥ 18 years old at time of screening
2. Subject has a clinical diagnosis of Type 1 diabetes for ≥ 2 years prior to screening as determined via source documentation
3. On MDI therapy (defined as ≥ 3 insulin injections per day and/or a basal/bolus regimen) ≥ 2 years prior to screening
4. Subject has been followed and treated by the investigator at this investigational site for at least 3 months prior to screening and subject has already undergone local educational therapeutic programs.
5. Subject is using:

   * Flash Glucose Monitoring (FGM) for ≥ 3 months with a daily average number of scans ≥ 5 over and with sensor readings > 70% of time over the previous month prior to screening (based on sensor usage from the download summary report of the FGM system over 30 days prior to screening) Or
   * Continuous Glucose Monitoring (CGM) for ≥ 3 months with a frequency of sensor use ≥ 70% of the time over the previous month prior to screening (based on download summary report from the CGM system over 30 days prior to screening).
6. Subject has a glycosylated hemoglobin (HbA1c) ≥ 8.0% (64 mmol/mol) at time of screening visit (as processed by a Central Lab).
7. Subject is willing to take or switch to one of the following insulins:

   1. Humalog™ (insulin lispro injection)
   2. NovoLog™ (insulin aspart)
8. Subject must have a minimum daily insulin requirement (Total Daily Dose) of ≥ 8 units and a maximum of 250 units.
9. Subject is willing to upload data from the study pump and meter, must have Internet access and a compatible computer system that meets the requirements for uploading the study pump data at home.
10. Subject is willing and able to sign and date informed consent, comply with all study procedures and wear all study devices, as required during the study.

Exclusion Criteria:

1. Subject has untreated Addison's disease, thyroid disorder, growth hormone deficiency, hypopituitarism or definite gastroparesis, per investigator judgment.
2. Subject is using pramlintide, DPP-4 inhibitor, GLP-1 agonists/mimetics, metformin, SGLT2 inhibitors at time of screening.
3. Subject has had renal failure defined by creatinine clearance <30 ml/min, as assessed by local lab test ≤ 12 months before screening or performed at screening at local lab, as defined by the creatinine-based Cockcroft or MDRD equations.
4. Subject is planning to switch from FGM to CGM therapy during the 6 months study phase. Note: Subject randomized to Control Arm should remain on their current FGM or CGM therapy during the study phase and will be switched to AHCL during the continuation phase.
5. Subject has a history of hearing or vision impairment hindering perception of glucose display and alarms, or otherwise incapable of using the study devices, per investigator judgment.
6. Women of child-bearing potential who have a positive pregnancy test at screening or plan to become pregnant during the course of the study.
7. Females who are sexually active and able to conceive will be excluded if they are not using an effective method of contraception and do not agree to continue using an effective method of contraception for the duration of the study, per investigator judgment.
8. Subject has any unresolved adverse skin conditions in the area of sensor placement (e.g. psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
9. Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or device in the last 2 weeks before enrollment into this study, as per investigator judgment.
10. Subject is currently abusing illicit drugs, marijuana, alcohol or prescription drugs (other than nicotine), per investigator judgment.
11. Subject has any other disease or condition that may preclude the patient from participating in the study, per investigator judgment.
12. Subject is legally incompetent, illiterate or vulnerable person.
13. Research staff involved with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2022-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- France (6):
  - Centre Hospitalier Universitaire Besancon - Hôpital Jean Minjoz, Besançon
  - CHU de Bordeaux - Hôpital Saint André, Bordeaux
  - CHU Caen, Caen
  - Hospices Civils de Lyon (DIAB-e CARE), Lyon
  - APM - Hôpital de la Conception, Marseille
  - Hospital Civil, Strasbourg
- Germany (4):
  - Diabetologische Schwerpunktpraxis Dr. Ralf Kolassa, Bergheim
  - Zentrum für Diabetologie Bergedorf, Hamburg
  - Gemeinschaftspraxis im Westtor Hausarztpraxis & Diabetologische Schwerpunktpraxis, Lage
  - Medical Center am Clemenshospital Dr. Winfried Keuthage, Münster
- United Kingdom (4):
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrooke's Hospital, Cambridge
  - Harrogate and District Hospital - NHS Foundation Trust, Harrogate
  - University Hospitals of Leicester NHS Trust Leicester General Hospital, Leicester
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jendle J, Buompensiere MI, Ozdemir Saltik AZ, de Portu S, Smith-Palmer J, Pollock RF, Cohen O. A European Cost-Utility Analysis of the MiniMed 780G Advanced Hybrid Closed-Loop System Versus Intermittently Scanned Continuous Glucose Monitoring with Multiple Daily Insulin Injections in People Living with Type 1 Diabetes. Diabetes Technol Ther. 2023 Dec;25(12):864-876. doi: 10.1089/dia.2023.0297. PMID 37801658
- [Derived] Edd SN, Castaneda J, Choudhary P, Kolassa R, Keuthage W, Kroeger J, Thivolet C, Evans M, Re R, Cellot J, de Portu S, Vorrink L, Shin J, van den Heuvel T, Cohen O; ADAPT study Group. Twelve-month results of the ADAPT randomized controlled trial: Reproducibility and sustainability of advanced hybrid closed-loop therapy outcomes versus conventional therapy in adults with type 1 diabetes. Diabetes Obes Metab. 2023 Nov;25(11):3212-3222. doi: 10.1111/dom.15217. Epub 2023 Aug 8. PMID 37551542
- [Derived] Choudhary P, Kolassa R, Keuthage W, Kroeger J, Thivolet C, Evans M, Re R, de Portu S, Vorrink L, Shin J, Habteab A, Castaneda J, da Silva J, Cohen O; ADAPT study Group. Advanced hybrid closed loop therapy versus conventional treatment in adults with type 1 diabetes (ADAPT): a randomised controlled study. Lancet Diabetes Endocrinol. 2022 Oct;10(10):720-731. doi: 10.1016/S2213-8587(22)00212-1. Epub 2022 Sep 1. PMID 36058207
- [Derived] de Portu S, Vorrink L, Re R, Shin J, Castaneda J, Habteab A, Cohen O. Randomised controlled trial of Advanced Hybrid Closed Loop in an Adult Population with Type 1 Diabetes (ADAPT): study protocol and rationale. BMJ Open. 2022 Feb 2;12(2):e050635. doi: 10.1136/bmjopen-2021-050635. PMID 35110310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first subject enrollment: 13-JUL-2020, Date of last subject visit (of study phase): 02-DEC-2021 Date of last subject visit (of continuation phase): 30-MAY-2022
Pre-assignment Details: 122 adults with type 1 diabetes consented to participate in the study. Of them, 19 subjects are Screen Failure. After 8 patients early exited before randomization, 95 (82 in Cohort A, 13 in Cohort B) subjects were randomized in study phase.
Groups:
- Cohort A - Treatment Arm: In study phase, subjects on MDI with Flash Glucose Monitoring (FGM) in run-in phase started using AHCL (stop MDI + FGM therapy at Visit 6A).
  In continuation phase, subjects continued using AHCL.
- Cohort A - Control Arm: In study phase, subjects on MDI with Flash Glucose Monitoring (FGM) in run-in phase continued using MDI + FGM.
  In continuation phase, subjects started using AHCL.
- Cohort B - Treatment Arm: In study phase, subjects on MDI + Real-Time CGM in run-in phase started using AHCL (stop MDI + CGM therapy at Visit 6A).
  In continuation phase, subjects continued using AHCL.
- Cohort B - Control Arm: In study phase, subjects on MDI + Real-Time CGM in run-in phase continued using MDI + CGM.
  In continuation phase, subjects started using AHCL.
Period: Study Phase
Arm/Group | Cohort A - Treatment Arm | Cohort A - Control Arm | Cohort B - Treatment Arm | Cohort B - Control Arm
Started | 41 (Subjects entering the study phase (randomized)) | 41 (Subjects entering the study phase (randomized)) | 8 (Subjects entering the study phase (randomized)) | 5 (Subjects entering the study phase (randomized))
Completed | 36 | 39 | 8 | 5
Not Completed | 5 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 2 | 0 | 0
Period: Continuation Phase
Arm/Group | Cohort A - Treatment Arm | Cohort A - Control Arm | Cohort B - Treatment Arm | Cohort B - Control Arm
Started | 36 | 39 (One subject in cohort A control arm withdrew at day of completion of study phase) | 8 | 5
Completed | 35 | 32 | 7 | 5
Not Completed | 1 | 7 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Subjects Randomized to Corresponding Group
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - Treatment Arm | Cohort A - Control Arm | Cohort B - Treatment Arm | Cohort B - Control Arm | Total
Number analyzed (Participants) | 41 | 41 | 8 | 5 | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.5 (11.63) | 39.7 (13.12) | 45.4 (13.32) | 36.2 (15.80) | 40.7 (12.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 16 | 3 | 3 | 44
  Male | 19 | 25 | 5 | 2 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
HbA1c [Mean (Standard Deviation); unit: Percentage] | 9.00 (0.972) | 9.07 (0.716) | 8.90 (0.457) | 9.46 (0.611) | 9.05 (0.815)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c 6 Months Change Between AHCL and MDI
Description: The difference in the mean HbA1c change (6 months - baseline) between the AHCL and the MDI + FGM arm will be evaluated (Cohort A).
Time Frame: Baseline and end of 6-month study phase
Population: Study phase: 82 subjects in Cohort A. 74 subjects have available measurements.
Measure: Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Cohort A - Treatment Arm | Cohort A - Control Arm
Number analyzed (Participants) | 36 | 38
Percentage of HbA1c | -1.54 (0.729) | -0.20 (0.797)
Statistical Analysis 1: Comparison: Cohort A - Treatment Arm vs Cohort A - Control Arm; Test type: Superiority; p < 0.0001, linear mixed model; Mean Difference (Final Values) = -1.42, 95% CI 2-sided [-1.74 to -1.10]

2. Secondary Outcome: TIR Between 70-180 mg/dL
Description: % Time spent within range with sensor glucose (SG) between 70 - 180 mg/dL (3.9-10.0 mmol/L). The difference in the mean between the AHCL and the MDI + FGM arm will be evaluated (Cohort A).
Time Frame: 6 months study phase
Population: Study phase: 82 subjects in Cohort A. 67 subjects have available measurements.
Measure: Mean (Standard Error); unit: Percentage of Time
Arm/Group | Cohort A - Treatment Arm | Cohort A - Control Arm
Number analyzed (Participants) | 36 | 31
Percentage of Time | 70.63 (9.700) | 43.59 (15.369)
Statistical Analysis 1: Comparison: Cohort A - Treatment Arm vs Cohort A - Control Arm; Test type: Superiority; p < 0.0001, linear mixed model; Mean Difference (Final Values) = 27.59, 95% CI 2-sided [21.59 to 33.60]

3. Secondary Outcome: Time in Hyperglycemic Range
Description: % Time spent in hyperglycemic range with SG > 180 mg/dL (> 10.0 mmol/L). The difference in the mean between the AHCL and the MDI + FGM arm will be evaluated (Cohort A).
Time Frame: 6 months study phase
Population: Study phase: 82 subjects in Cohort A. 67 subjects have available measurements.
Measure: Mean (Standard Error); unit: Percentage of Time
Arm/Group | Cohort A - Treatment Arm | Cohort A - Control Arm
Number analyzed (Participants) | 36 | 31
Percentage of Time | 26.74 (10.444) | 53.81 (16.465)
Statistical Analysis 1: Comparison: Cohort A - Treatment Arm vs Cohort A - Control Arm; Test type: Superiority; p < 0.0001, linear mixed model; Mean Difference (Final Values) = -27.86, 95% CI 2-sided [-34.16 to -21.55]

4. Secondary Outcome: Hypoglycemic Events
Description: Number of biochemical hypoglycemic events< 54 mg/dL (3.0 mmol/L) (defined as sensor values < 54 mg/dL (3.0 mmol/L) per 15 consecutive minutes (Danne, 2017). When the time between two successive events is less than 30 minutes, they will be combined and counted as one event. The difference in the mean between the AHCL and the MDI + FGM arm will be evaluated (Cohort A)
Time Frame: 6 months study phase
Population: Study phase: 82 subjects in Cohort A. 67 subjects have available measurements.
Measure: Mean (Standard Error); unit: Events per week
Arm/Group | Cohort A - Treatment Arm | Cohort A - Control Arm
Number analyzed (Participants) | 36 | 31
Events per week | 1.29 (1.322) | 0.98 (1.436)
Statistical Analysis 1: Comparison: Cohort A - Treatment Arm vs Cohort A - Control Arm; Test type: Superiority; p = 0.6227, linear mixed model; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.37 to 0.61]

5. Other Pre Specified Outcome: HbA1c 6 Months Change Between AHCL and MDI
Description: The difference in the mean HbA1c change (6 months - baseline) between the AHCL and the MDI + CGM arm will be evaluated (Cohort B).
Time Frame: Baseline and end of 6-month study phase
Population: Study phase: 13 subjects in Cohort B. 12 subjects have available measurements.
Measure: Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Cohort B - Treatment Arm | Cohort B - Control Arm
Number analyzed (Participants) | 7 | 5
Percentage of HbA1c | -1.70 (1.039) | -0.60 (1.259)
Statistical Analysis 1: Comparison: Cohort B - Treatment Arm vs Cohort B - Control Arm; Test type: Superiority; linear mixed model — Due to the small sample size, p value will not be meaningful. Therefore, p value is not presented; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-2.17 to 0.00]

6. Other Pre Specified Outcome: TIR Between 70-180 mg/dL
Description: % Time spent within range with sensor glucose (SG) between 70 - 180 mg/dL (3.9-10.0 mmol/L). The difference in the mean between the AHCL and the MDI + CGM arm will be evaluated (Cohort B).
Time Frame: 6 months study phase
Population: Study phase: 13 subjects in Cohort B. 13 subjects have available measurements.
Measure: Mean (Standard Error); unit: Percentage of Time
Arm/Group | Cohort B - Treatment Arm | Cohort B - Control Arm
Number analyzed (Participants) | 8 | 5
Percentage of Time | 73.63 (13.749) | 46.41 (12.547)
Statistical Analysis 1: Comparison: Cohort B - Treatment Arm vs Cohort B - Control Arm; Test type: Superiority; linear mixed model — Due to the small sample size, p value will not be meaningful. Therefore, p value is not presented; Mean Difference (Final Values) = 28.81, 95% CI 2-sided [12.34 to 45.28]

7. Other Pre Specified Outcome: Time in Hyperglycemic Range
Description: % Time spent in hyperglycemic range with SG > 180 mg/dL (> 10.0 mmol/L). The difference in the mean between the AHCL and the MDI + CGM arm will be evaluated (Cohort B).
Time Frame: 6 months study phase
Population: Study phase: 13 subjects in Cohort B. 13 subjects have available measurements.
Measure: Mean (Standard Error); unit: Percentage of Time
Arm/Group | Cohort B - Treatment Arm | Cohort B - Control Arm
Number analyzed (Participants) | 8 | 5
Percentage of Time | 23.97 (13.512) | 50.88 (15.630)
Statistical Analysis 1: Comparison: Cohort B - Treatment Arm vs Cohort B - Control Arm; Test type: Superiority; linear mixed model — Due to the small sample size, p value will not be meaningful. Therefore, p value is not presented; Mean Difference (Final Values) = -28.45, 95% CI 2-sided [-45.27 to -11.64]

8. Other Pre Specified Outcome: Hypoglycemic Events
Description: Number of biochemical hypoglycemic events< 54 mg/dL (3.0 mmol/L) (defined as sensor values < 54 mg/dL (3.0 mmol/L) per 15 consecutive minutes (Danne, 2017). When the time between two successive events is less than 30 minutes, they will be combined and counted as one event. The difference in the mean between the AHCL and the MDI + CGM arm will be evaluated (Cohort B).
Time Frame: 6 months study phase
Population: Study phase: 13 subjects in Cohort B. 13 subjects have available measurements.
Measure: Mean (Standard Error); unit: Events per week
Arm/Group | Cohort B - Treatment Arm | Cohort B - Control Arm
Number analyzed (Participants) | 8 | 5
Events per week | 1.07 (1.327) | 0.93 (1.135)
Statistical Analysis 1: Comparison: Cohort B - Treatment Arm vs Cohort B - Control Arm; Test type: Superiority; linear mixed model — Due to the small sample size, p value will not be meaningful. Therefore, p value is not presented; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-1.32 to 0.59]

9. Other Pre Specified Outcome: HbA1c 6 Months Change Within Group
Description: The change in the mean HbA1c from end of 6-month study phase to end of 6-month continuation phase will be evaluated (Cohort A)
Time Frame: End of 6-month study phase and end of 6-month continuation phase
Population: Continuation phase: 36 subjects in Cohort A Treatment Arm. 33 subjects have available measurements.
Measure: Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Cohort A - Treatment Arm
Number analyzed (Participants) | 33
Percentage of HbA1c | 0.16 (0.491)

10. Other Pre Specified Outcome: HbA1c 6 Months Change Within Group
Description: as for outcome 9
Time Frame: End of 6-month study phase and end of 6-month continuation phase
Description (as registered): The change in the mean HbA1c from end of 6-month study phase to end of 6-month continuation phase will be evaluated (Cohort B).
Population: Continuation phase: 38 subjects in Cohort A Control Arm. 31 subjects have available measurements.
Measure: Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Cohort A - Control Arm
Number analyzed (Participants) | 31
Percentage of HbA1c | -1.36 (0.777)

11. Other Pre Specified Outcome: HbA1c 12 Months Change Between Groups
Description: The difference in the mean HbA1c change (12 months - baseline) between treatment arm and control arm will be evaluated (Cohort A)
Time Frame: Baseline through the end of 6-month continuation phase (a total of 12 months)
Population: Overall study: 82 subjects in Cohort A. 66 subjects have available measurements.
Measure: Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Cohort A - Treatment Arm | Cohort A - Control Arm
Number analyzed (Participants) | 34 | 32
Percentage of HbA1c | -1.47 (0.829) | -1.58 (0.828)

12. Other Pre Specified Outcome: HbA1c 6 Months Change Within Group
Description: The change in the mean HbA1c from end of 6-month study phase to end of 6-month continuation phase will be evaluated (Cohort B).
Time Frame: End of 6-month study phase and end of 6-month continuation phase
Population: Continuation phase: 8 subjects in Cohort B Treatment Arm. 5 subjects have available measurements.
Measure: Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Cohort B - Treatment Arm
Number analyzed (Participants) | 5
Percentage of HbA1c | 0.02 (0.466)

13. Other Pre Specified Outcome: HbA1c 6 Months Change Within Group
Description: as for outcome 12
Time Frame: End of 6-month study phase and end of 6-month continuation phase
Population: Continuation phase: 5 subjects in Cohort B Control Arm. 3 subjects have available measurements.
Measure: Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Cohort B - Control Arm
Number analyzed (Participants) | 3
Percentage of HbA1c | -0.67 (0.551)

14. Other Pre Specified Outcome: HbA1c 12 Months Change Between Groups
Description: The difference in the mean HbA1c change (12 months - baseline) between treatment arm and control arm will be evaluated (Cohort B).
Time Frame: Baseline through the end of 6-month continuation phase (a total of 12 months).
Population: Overall study: 13 subjects in Cohort B. 9 subjects have available measurements.
Measure: Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Cohort B - Treatment Arm | Cohort B - Control Arm
Number analyzed (Participants) | 6 | 3
Percentage of HbA1c | -1.33 (1.122) | -1.30 (0.529)

ADVERSE EVENTS:
Time Frame: 4 weeks of Run-in Phase, 6 months of Study Phase, 6 months of Continuation Phase
Groups:
- Cohort A Run-in Phase: Subjects were using MDI with Flash Glucose Monitoring (FGM).
- Cohort B Run-in Phase: Subjects were using MDI + Real-Time CGM.
- Cohort A - Treatment Arm Study Phase: In study phase, subjects on MDI with Flash Glucose Monitoring (FGM) in run-in phase started using AHCL (stop MDI + FGM therapy at Visit 6A).
- Cohort A - Control Arm Study Phase: In study phase, subjects on MDI with Flash Glucose Monitoring (FGM) in run-in phase continued using MDI + FGM.
- Cohort B - Treatment Arm Study Phase: In study phase, subjects on MDI + Real-Time CGM in run-in phase started using AHCL (stop MDI + CGM therapy at Visit 6A).
- Cohort B - Control Arm Study Phase: In study phase, subjects on MDI + Real-Time CGM in run-in phase continued using MDI + CGM.
- All Patients Continuation Phase: All subjects were using AHCL in continuation phase.
Arm/Group | Cohort A Run-in Phase | Cohort B Run-in Phase | Cohort A - Treatment Arm Study Phase | Cohort A - Control Arm Study Phase | Cohort B - Treatment Arm Study Phase | Cohort B - Control Arm Study Phase | All Patients Continuation Phase
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/17 | 0/41 | 0/41 | 0/8 | 0/5 | 0/88
Serious Adverse Events (participants affected / at risk) | 1/105 | 1/17 | 1/41 | 1/41 | 1/8 | 0/5 | 2/88
Other Adverse Events (participants affected / at risk) | 21/105 | 1/17 | 19/41 | 18/41 | 2/8 | 0/5 | 31/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Run-in Phase (N=105) | Cohort B Run-in Phase (N=17) | Cohort A - Treatment Arm Study Phase (N=41) | Cohort A - Control Arm Study Phase (N=41) | Cohort B - Treatment Arm Study Phase (N=8) | Cohort B - Control Arm Study Phase (N=5) | All Patients Continuation Phase (N=88)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Run-in Phase (N=105) | Cohort B Run-in Phase (N=17) | Cohort A - Treatment Arm Study Phase (N=41) | Cohort A - Control Arm Study Phase (N=41) | Cohort B - Treatment Arm Study Phase (N=8) | Cohort B - Control Arm Study Phase (N=5) | All Patients Continuation Phase (N=88)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal weight gain (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 8 (9)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Catheter site mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 4 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immunisation reaction (Immune system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Medical device site bruise (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site haemorrhage (General disorders) | 5 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Medical device site irritation (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Medical device site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Medical device site reaction (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Open angle glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polycystic ovaries (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT04235504/Prot_000.pdf
  • Statistical Analysis Plan: Study Phase (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT04235504/SAP_001.pdf
  • Statistical Analysis Plan: Continuation Phase (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT04235504/SAP_002.pdf